CLINICAL TRIAL: NCT06945575
Title: Comparison of T-loop vs Opus Loop in Canine Retraction Efficacy and Anchorage Loss Control - a Split- Mouth, Randomized Clinical Trial
Brief Title: Comparison of T-loop vs Opus Loop in Canine Retraction Efficacy and Anchorage Loss Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Maria Moin, Assistant professor, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DowUHS 2
Record Dates: First submitted 2025-03-17; First posted 2025-04-25 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-04

CONDITIONS: Space Closure, Orthodontic
MeSH Terms: interventions — Opus PCF

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Opus loop (Active Comparator): Opus loop will be inserted from 1st molar to canine for canine retraction. it will be activated every month
  Interventions: Other: Opus loop
- T-loop (Active Comparator): T loop will be inserted from 1st molar to canine for canine retraction. it will be activated every month
  Interventions: Other: T loop

INTERVENTIONS:
Other: Opus loop — 17X25SS will used to fabricate opus loop which is L shaped loop with helix
  Other Names: opus
  Arms: Opus loop
Other: T loop — 17X25SS wire will be used to fabricate T-loop which is a T shaped loop
  Arms: T-loop

SUMMARY:
The primary aim of this split-mouth randomized control trial is to compare the rate of canine retraction between the T loop and the Opus loop. The secondary objectives are to compare the angulation of the canine, changes in the first molar position in terms of anchorage loss, and molar rotation for the two loops used T-loop and Opus loop will be placed randomly on the right and left quadrants of patients for canine retraction and outcomes will be measured before and after completion of canine retraction

DETAILED DESCRIPTION:
T-loop and Opus loop will be placed in the right and left quadrants of the patient for canine retraction after initial leveling and alignment. canine retraction rate will be measured by using a calibrated caliper every month. canine angulation will be evaluated by periapical x-ray which will be taken before and after completion of canine retraction and anchorage loss and molar rotation will be assessed by model analysis

ELIGIBILITY:
Inclusion Criteria:

Age between 14 -40 years Extractions of maxillary 1st premolars Class 1, 1/4th, 1/2, and 3/4th unit Class II molar relation Presence of all teeth up to the second molar Good oral hygiene

Exclusion Criteria:

Full cusp Class II Developmental, medical, or genetic problems Patient using bisphosphonates Spacing in dentition Grossly carious upper molars that cannot be restored Patient with active periodontal disease Severe crowding

Ages: 14 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2025-02-04 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Rate of canine retraction | From enrollment till end of treatment at 4 months
  The rate of canine retraction will be calculated by "the amount of canine retraction (in millimeters) divided by the time interval". The amount of canine retraction will be assessed by measuring the distance from the canine cusp tip to the mesio-buccal (MB) cusp tip of the 1st molar with a calibrated caliper at the time of placement of loops and at every month by a single calibrated clinician. The duration will be measured as a time interval and each time interval will be 4 weeks.

SECONDARY OUTCOMES:
Change in canine angulation at start of canine retraction and at the end of canine retraction | From enrollment till end of treatment at 4 months
  DIGORA™ Optime will be used take periapical radiographs of maxillary canine to 1st molar at the start of canine retraction and after completion of canine retraction. X-ray film holders will be used while taking periapical radiographs for standardization of X-rays. A single calibrated examiner will analyse angulation of canine by measuring an angle between vertical line drawn from buccal cusp tip of canine till root apex in reference with 2nd premolar using a protractor.
Change in anchorage loss before and after completion of canine retraction | From enrollment till end of treatment at 4 months
  A dental cast will be made by taking an alginate impression of the patient. Anchorage loss will be measured by drawing a horizontal line from the mesiobuccal cusp tip of the right and left 1st molars. The distance between the 3rd rugae and this horizontal line will be measured on both sides using a millimetric scale, and the difference between the distance at start and after completion of canine retraction will be measured as anchorage loss.
Change in molar rotation at before and after completion of canine reatraction | From enrollment till end of treatment at 4 months
  dental cast will be evaluated before and after canine retraction. A diagonal line will be drawn from both left and right 1st molar distobuccal cusp tip to mesiopalatal cusp tip till mid palatal raphe. The angle formed between diagonal line and mid midpalatal raphe will be measured from both the left and right sides using a protractor. The difference between angle before and after canine retraction will be measured as a change in molar rotation

CONTACTS AND LOCATIONS:
Locations (1):
- Bahria University Health Sciences, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided